CLINICAL TRIAL: NCT00225082
Title: SNAP: Switching Nucleoside Analogues Protocol - Lipoatrophy and Mitochondrial
Brief Title: SNAP: Switching Nucleoside Analogues Protocol - Lipoatrophy and Mitochondrial Function
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Robert Murphy, MD, Northwestern University
Other Study IDs: SNAP
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection
Keywords: Lipoatrophy; Mitochondrial function; Nucleoside analogue switch; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — adipose tissue, blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nucleoside analogue switch — stavudine switched to tenofovir

SUMMARY:
HIV infected subjects receiving antiretroviral treatment for greater than 6 years with be evaluated for clinical lipoatrophy and mitochondrial function after switching nucleoside analogues from stavudine (d4T) to tenofovir treatment and after 4.

Hypothesis: Tenofovir therapy will increase peripheral fat content as assessed by DEXA and mitochondrial function at 48 weeks.

DETAILED DESCRIPTION:
HIV infected subjects receiving antiretroviral treatment (lopinavir/ritonavir, stavudine, and lamivudine) for greater than 6 years through the Abbott M97-720 protocol with be evaluated for clinical lipoatrophy and mitochondrial function prior to switching nucleoside analogues from stavudine (d4T) to tenofovir and after 48 weeks or tenofovir treatment.

Subjects with or without lipoatrophy are eligible for the study. Adipose tissue biopsies to measure mitochondrial function, metabolic laboratory tests, and DAXA scans and clinical evaluations of lipodystrophy will be performed at Entry and after 48 weeks of tenofovir treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Receiving Kaletra, stavudine, and lamivudine for greater than 6 years (through Abbott M97-720 study)
* Planning to switch from stavudine to tenofovir

Exclusion Criteria:

* Will continue to receive stavudine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected subjects receiving antiretroviral treatment (lopinavir/ritonavir, stavudine, and lamivudine) for greater than 6 years through the Abbott M97-720 protocol with be evaluated for clinical lipoatrophy and mitochondrial function prior to switching nucleoside analogues from stavudine (d4T) to tenofovir and after 48 weeks or tenofovir treatment. Subjects with or without lipoatrophy are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2004-11; Primary Completion 2006-12 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Murphy, MD, Study Chair — Northwestern University; Mariana Gerschenson, Ph.D., Study Chair — University of Hawaii
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Gerschenson M, Kim C, Berzins B, Taiwo B, Libutti DE, Choi J, Chen D, Weinstein J, Shore J, da Silva B, Belsey E, McComsey GA, Murphy RL. Mitochondrial function, morphology and metabolic parameters improve after switching from stavudine to a tenofovir-containing regimen. J Antimicrob Chemother. 2009 Jun;63(6):1244-50. doi: 10.1093/jac/dkp100. Epub 2009 Mar 25. PMID 19321503